CLINICAL TRIAL: NCT01597258
Title: SPECIAL INVESTIGATION OF XALKORI FOR NSCLC (REGULATORY POST MARKETING COMMITMENT PLAN)
Brief Title: Safety And Efficacy Of Crizotinib (Regulatory Post Marketing Commitment Plan)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A8081031
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Safety; All cases surveillance in Japan; ALK-positive unresectable advanced and/or recurrent non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Crizotinib (Xalkori)
  Interventions: Drug: Crizotinib (Xalkori)

INTERVENTIONS:
Drug: Crizotinib (Xalkori) — XALKORI® Capsule 200 mg／XALKORI® Capsule 250 mg This surveillance is all cases surveillance based on Japanese regulation. Frequency and duration are according to Package Insert as follows. " The recommended dose schedule of crizotinib is 250 mg taken orally twice daily. Dosing interruption and/or dose reduction may be required based on patients' clinical status. "
  Other Names: XALKORI® Capsule 200 mg／XALKORI® Capsule 250 mg

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes Crizotinib (XALKORI) should be registered.

ELIGIBILITY:
Inclusion Criteria:

* All the patients whom an investigator prescribes XALKORI. (Patients need to be administered Crizotinib (XALKORI) in order to be enrolled in this all cases surveillance.)

Exclusion Criteria:

* Patients not administered XALKORI in spite of enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients whom an investigator involving A8081031 prescribes the Crizotinib (XALKORI).
Sampling Method: Probability Sample
Enrollment: 2029 (Actual)
Dates: Start 2012-05-29 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Ueno N, Banno S, Endo Y, Tamura M, Sugaya K, Hashigaki S, Ohki E, Yoshimura A, Gemma A. Treatment status and safety of crizotinib in 2028 Japanese patients with ALK-positive NSCLC in clinical settings. Jpn J Clin Oncol. 2019 Jul 1;49(7):676-686. doi: 10.1093/jjco/hyz049. PMID 31008509
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081031&StudyName=Safety%20And%20Efficacy%20Of%20Crizotinib%20%28Regulatory%20Post%20Marketing%20Commitment%20Plan%29

RESULTS

PARTICIPANT FLOW:
Groups:
- XALKORI Capsules (Crizotinib): Participants who received XALKORI Capsules as indicated in the approved local product document were observed for a period of 52 weeks. The dosage can be adjusted as per physician's discretion.
Period: Overall Study
Arm/Group | XALKORI Capsules (Crizotinib)
Started | 2029
Completed | 2028
Not Completed | 1
Not completed — No Drug Administration | 1

BASELINE CHARACTERISTICS:
Population: A total of 2029 participants were completed this study. Of the 2029 participants, 1 participant was excluded from the safety analysis set due to no drug administration.
Arm/Group | XALKORI Capsules (Crizotinib)
Number analyzed (Participants) | 2028
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 1221
  ≥65 years | 803
  Unknown | 4
Sex/Gender, Customized [Number; unit: Participants]
  Male | 937
  Female | 1087
  Unknown | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Drug Reactions
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to XALKORI Capsules in a participant who received XALKORI Capsules. A serious ADR was a ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to XALKORI Capsules was assessed by the physician.
Time Frame: 52 weeks
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and had received XALKORI Capsules at least once.
Measure: Number; unit: Participants
Arm/Group | XALKORI Capsules (Crizotinib)
Number analyzed (Participants) | 2028
Participants
  ADR | 1858
  Serious ADR | 518

2. Secondary Outcome: Objective Response Rate (ORR) at 52 Weeks
Description: Clinical effectiveness of XALKORI Capsules was assessed as "complete response (CR)", "partial response (PR)", "stable disease (SD)", "progressive disease (PD)", or "indeterminate" by the physician, based on Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.1. Overall effectiveness of XALKORI Capsules was determined by the physician based on the best response. Clinical effectiveness rate was ORR, defined as the percentage of subjects achieving CR or PR with best response. The ORR was presented along with the corresponding exact 2-sided 95% confidence interval (CI).
Time Frame: 52 weeks
Population: The efficacy analysis set (EAS) is comprised in the safety analysis set who had at least one measurable lesion and were evaluated for effectiveness. 1633 participants were included in the EAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | XALKORI Capsules (Crizotinib)
Number analyzed (Participants) | 1633
Percentage of participants | 66.5 [64.2 to 68.8]

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | XALKORI Capsules (Crizotinib)
All-Cause Mortality (participants affected / at risk) | 436/2028
Serious Adverse Events (participants affected / at risk) | 777/2028
Other Adverse Events (participants affected / at risk) | 1783/2028
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XALKORI Capsules (Crizotinib) (N=2028)
Venous thrombosis limb (Vascular disorders) | 2
Vena cava thrombosis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Peripheral circulatory failure (Vascular disorders) | 1
Hypotension (Vascular disorders) | 4
Embolism venous (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 10
Circulatory collapse (Vascular disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 22
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 11
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 7
Renal disorder (Renal and urinary disorders) | 3
Renal cyst (Renal and urinary disorders) | 4
Neurogenic bladder (Renal and urinary disorders) | 1
Bladder disorder (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Suicide attempt (Psychiatric disorders) | 3
Major depression (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 5
Completed suicide (Psychiatric disorders) | 1
Syncope (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 6
Presyncope (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Paraneoplastic neurological syndrome (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 3
Neuralgia (Nervous system disorders) | 1
Myasthenia gravis (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Guillain-Barre syndrome (Nervous system disorders) | 1
Facial paralysis (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 2
Encephalopathy (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Dysarthria (Nervous system disorders) | 1
Drug withdrawal convulsions (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Depressed level of consciousness (Nervous system disorders) | 7
Cerebellar infarction (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 4
Altered state of consciousness (Nervous system disorders) | 2
Akathisia (Nervous system disorders) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 293
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaplastic large-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 19
White blood cell count increased (Investigations) | 1
White blood cell count decreased (Investigations) | 5
Weight increased (Investigations) | 1
Renal function test abnormal (Investigations) | 1
Platelet count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 22
Hepatic enzyme increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Eosinophil count increased (Investigations) | 1
Electrocardiogram T wave abnormal (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 10
C-reactive protein increased (Investigations) | 3
Blood creatinine increased (Investigations) | 12
Blood creatine phosphokinase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood albumin decreased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 22
Alanine aminotransferase increased (Investigations) | 22
Spinal fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Compression fracture (Injury, poisoning and procedural complications) | 1
Wound infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 5
Sepsis (Infections and infestations) | 5
Renal cyst infection (Infections and infestations) | 2
Renal abscess (Infections and infestations) | 12
Pyelonephritis acute (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Psoas abscess (Infections and infestations) | 2
Pseudomembranous colitis (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 3
Pneumonia influenzal (Infections and infestations) | 1
Pneumonia herpes viral (Infections and infestations) | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 12
Pneumonia (Infections and infestations) | 45
Pneumocystis jirovecii pneumonia (Infections and infestations) | 5
Peritonitis (Infections and infestations) | 2
Perinephric abscess (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 3
Muscle abscess (Infections and infestations) | 1
Mediastinitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 5
Lung abscess (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 2
Kidney infection (Infections and infestations) | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 3
Infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Gastroenteritis salmonella (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Abdominal abscess (Infections and infestations) | 1
Liver disorder (Hepatobiliary disorders) | 15
Hepatotoxicity (Hepatobiliary disorders) | 18
Hepatitis fulminant (Hepatobiliary disorders) | 2
Hepatitis acute (Hepatobiliary disorders) | 2
Hepatic necrosis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 52
Hepatic failure (Hepatobiliary disorders) | 2
Drug-induced liver injury (Hepatobiliary disorders) | 5
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Biliary dilatation (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Sudden death (General disorders) | 1
Pyrexia (General disorders) | 12
Pain (General disorders) | 1
Oedema peripheral (General disorders) | 4
Oedema (General disorders) | 8
Multiple organ dysfunction syndrome (General disorders) | 1
Malaise (General disorders) | 5
General physical health deterioration (General disorders) | 1
Face oedema (General disorders) | 1
Drug interaction (General disorders) | 1
Death (General disorders) | 5
Asthenia (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 37
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 16
Oesophageal ulcer (Gastrointestinal disorders) | 7
Oesophageal perforation (Gastrointestinal disorders) | 1
Oesophageal pain (Gastrointestinal disorders) | 1
Oesophageal fistula (Gastrointestinal disorders) | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1
Necrotising oesophagitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 34
Large intestine perforation (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 3
Ileus (Gastrointestinal disorders) | 4
Haematemesis (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal toxicity (Gastrointestinal disorders) | 1
Gastrointestinal oedema (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 1
Visual impairment (Eye disorders) | 2
Vision blurred (Eye disorders) | 2
Photopsia (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Macular hole (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Eye disorder (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Cataract (Eye disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 4
Long QT syndrome (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 11
Cardiac arrest (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 7
Arrhythmia (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 12
Leukopenia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 9
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 84
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 5
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XALKORI Capsules (Crizotinib) (N=2028)
Dysgeusia (Nervous system disorders) | 339
Decreased appetite (Metabolism and nutrition disorders) | 210
White blood cell count decreased (Investigations) | 109
Blood creatinine increased (Investigations) | 190
Neutrophil count decreased (Investigations) | 166
Blood alkaline phosphatase increased (Investigations) | 115
Aspartate aminotransferase increased (Investigations) | 271
Alanine aminotransferase increased (Investigations) | 291
Liver disorder (Hepatobiliary disorders) | 145
Hepatic function abnormal (Hepatobiliary disorders) | 249
Pyrexia (General disorders) | 118
Oedema peripheral (General disorders) | 118
Vomiting (Gastrointestinal disorders) | 326
Nausea (Gastrointestinal disorders) | 633
Diarrhoea (Gastrointestinal disorders) | 500
Constipation (Gastrointestinal disorders) | 299
Visual impairment (Eye disorders) | 195
Photopsia (Eye disorders) | 384
Anaemia (Blood and lymphatic system disorders) | 78
Coagulopathy (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Leukocytosis (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 14
Lymphadenitis (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 45
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Bradycardia (Cardiac disorders) | 90
Cardiac failure (Cardiac disorders) | 3
Cardiac tamponade (Cardiac disorders) | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1
Conduction disorder (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 5
Pericardial effusion (Cardiac disorders) | 3
Pericarditis (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 34
Tachycardia (Cardiac disorders) | 2
Ventricular arrhythmia (Cardiac disorders) | 1
Colour blindness (Congenital, familial and genetic disorders) | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1
Deafness (Ear and labyrinth disorders) | 2
Ear discomfort (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 4
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Abnormal sensation in eye (Eye disorders) | 1
Accommodation disorder (Eye disorders) | 1
Asthenopia (Eye disorders) | 1
Blepharitis (Eye disorders) | 1
Cataract (Eye disorders) | 2
Cataract subcapsular (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Diabetic retinopathy (Eye disorders) | 1
Diplopia (Eye disorders) | 87
Dry eye (Eye disorders) | 4
Extraocular muscle paresis (Eye disorders) | 1
Eye disorder (Eye disorders) | 6
Eyelid oedema (Eye disorders) | 2
Hypermetropia (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Night blindness (Eye disorders) | 2
Optic nerve disorder (Eye disorders) | 2
Periorbital oedema (Eye disorders) | 2
Photophobia (Eye disorders) | 54
Punctate keratitis (Eye disorders) | 1
Retinal tear (Eye disorders) | 1
Vision blurred (Eye disorders) | 85
Visual acuity reduced (Eye disorders) | 4
Vitreous floaters (Eye disorders) | 28
Abdominal discomfort (Gastrointestinal disorders) | 19
Abdominal distension (Gastrointestinal disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 24
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 29
Anal inflammation (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 5
Cheilitis (Gastrointestinal disorders) | 5
Chronic gastritis (Gastrointestinal disorders) | 2
Crohn's disease (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Dumping syndrome (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 12
Dysphagia (Gastrointestinal disorders) | 11
Enterocolitis (Gastrointestinal disorders) | 6
Epigastric discomfort (Gastrointestinal disorders) | 3
Faeces soft (Gastrointestinal disorders) | 10
Food poisoning (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 19
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 6
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 1
Gastrointestinal oedema (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 23
Glossodynia (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 4
Hiatus hernia (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 2
Intestinal dilatation (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Lip erosion (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 5
Oesophageal pain (Gastrointestinal disorders) | 6
Oesophageal stenosis (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 9
Oesophagitis (Gastrointestinal disorders) | 40
Oral dysaesthesia (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 1
Pancreatic cyst (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 34
Subileus (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 7
Chills (General disorders) | 1
Face oedema (General disorders) | 11
Fatigue (General disorders) | 18
Feeling abnormal (General disorders) | 1
Generalised oedema (General disorders) | 3
Infusion site extravasation (General disorders) | 2
Localised oedema (General disorders) | 3
Malaise (General disorders) | 93
Non-cardiac chest pain (General disorders) | 1
Oedema (General disorders) | 82
Pain (General disorders) | 11
Sensation of foreign body (General disorders) | 1
Thirst (General disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 6
Hepatic cyst (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 3
Hepatitis (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 69
Hypogammaglobulinaemia (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 4
Abscess oral (Infections and infestations) | 1
Angular cheilitis (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Atypical mycobacterial infection (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 23
Cellulitis (Infections and infestations) | 5
Conjunctivitis (Infections and infestations) | 4
Cystitis (Infections and infestations) | 12
Device related infection (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 2
Enterocolitis bacterial (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Gingivitis (Infections and infestations) | 3
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 13
Infection (Infections and infestations) | 6
Infectious pleural effusion (Infections and infestations) | 2
Influenza (Infections and infestations) | 3
Lower respiratory tract infection (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 2
Lung infection (Infections and infestations) | 13
Nasopharyngitis (Infections and infestations) | 23
Oesophageal candidiasis (Infections and infestations) | 9
Oral candidiasis (Infections and infestations) | 6
Oral herpes (Infections and infestations) | 4
Oropharyngeal candidiasis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 2
Otitis media acute (Infections and infestations) | 1
Paronychia (Infections and infestations) | 2
Parotitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 9
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 51
Pneumonia bacterial (Infections and infestations) | 6
Pulmonary tuberculosis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Skin candida (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Tinea infection (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 4
Tonsillitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 20
Chest injury (Injury, poisoning and procedural complications) | 1
Chillblains (Injury, poisoning and procedural complications) | 1
Closed globe injury (Injury, poisoning and procedural complications) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 2
Radiation pneumonitis (Injury, poisoning and procedural complications) | 11
Rib fracture (Injury, poisoning and procedural complications) | 2
Recall phenomenon (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 5
Tendon rupture (Injury, poisoning and procedural complications) | 1
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Amylase increased (Investigations) | 2
Beta 2 microglobulin increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 9
Blood calcium decreased (Investigations) | 1
Blood chloride decreased (Investigations) | 2
Blood chloride increased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 29
Blood lactate dehydrogenase increased (Investigations) | 23
Blood potassium increased (Investigations) | 5
Blood pressure decreased (Investigations) | 1
Blood urea abnormal (Investigations) | 1
Blood urea increased (Investigations) | 24
Carbohydrate antigen 19-9 increased (Investigations) | 1
Carcinoembryonic antigen increased (Investigations) | 3
Cardioactive drug level increased (Investigations) | 1
Cell marker increased (Investigations) | 2
Chest X-ray abnormal (Investigations) | 1
C-reactive protein increased (Investigations) | 11
Creatinine renal clearance decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 65
Gamma-glutamyltransferase increased (Investigations) | 9
Granulocyte count decreased (Investigations) | 1
Grip strength decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 9
Hepatic enzyme increased (Investigations) | 9
International normalised ratio increased (Investigations) | 3
Intraocular pressure increased (Investigations) | 2
Investigation abnormal (Investigations) | 1
Liver function test abnormal (Investigations) | 7
Liver function test increased (Investigations) | 9
Lymphocyte count decreased (Investigations) | 22
Lymphocyte count increased (Investigations) | 1
Monocyte count increased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Nutritional condition abnormal (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Platelet count decreased (Investigations) | 16
Platelet count increased (Investigations) | 4
Protein total decreased (Investigations) | 5
Prothrombin time prolonged (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
Renal function test abnormal (Investigations) | 1
Transaminases increased (Investigations) | 10
Tumour marker increased (Investigations) | 2
Vitamin B12 decreased (Investigations) | 1
Weight decreased (Investigations) | 5
Weight increased (Investigations) | 2
White blood cell count increased (Investigations) | 14
Blood albumin decreased (Investigations) | 5
Eosinophil count increased (Investigations) | 7
Glomerular filtration rate decreased (Investigations) | 2
Red blood cell count increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Fluid retention (Metabolism and nutrition disorders) | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 43
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 25
Hypocalcaemia (Metabolism and nutrition disorders) | 22
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 11
Hyponatraemia (Metabolism and nutrition disorders) | 15
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 3
Hypozincaemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Zinc deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 16
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 2
Amnesia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 55
Dizziness postural (Nervous system disorders) | 6
Dyslalia (Nervous system disorders) | 1
Facial neuralgia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 23
Hypoaesthesia (Nervous system disorders) | 21
Intracranial pressure increased (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
Muscle spasticity (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 7
Neuropathy peripheral (Nervous system disorders) | 28
Neurotoxicity (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 19
Pyramidal tract syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Sensory disturbance (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 8
Syncope (Nervous system disorders) | 2
Tension headache (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Trigeminal nerve disorder (Nervous system disorders) | 1
Visual field defect (Nervous system disorders) | 8
Visual perseveration (Nervous system disorders) | 77
Affective disorder (Psychiatric disorders) | 1
Anticipatory anxiety (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 4
Anxiety disorder (Psychiatric disorders) | 3
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 11
Depression (Psychiatric disorders) | 7
Dissociative disorder (Psychiatric disorders) | 1
Dysphoria (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 35
Mental disorder (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Neurosis (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Chromaturia (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 3
Glomerulonephritis chronic (Renal and urinary disorders) | 1
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 1
Nephropathy toxic (Renal and urinary disorders) | 3
Neurogenic bladder (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 1
Prerenal failure (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 3
Renal cyst (Renal and urinary disorders) | 12
Renal disorder (Renal and urinary disorders) | 22
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 73
Renal vein thrombosis (Renal and urinary disorders) | 1
Urethral stenosis (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 5
Amenorrhoea (Reproductive system and breast disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 26
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 16
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 25
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 24
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 24
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 7
Angioedema (Skin and subcutaneous tissue disorders) | 1
Asteatosis (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 11
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 12
Eczema (Skin and subcutaneous tissue disorders) | 11
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 6
Erythema annulare (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 18
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 19
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 59
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 3
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 7
Deep vein thrombosis (Vascular disorders) | 7
Embolism (Vascular disorders) | 3
Hypertension (Vascular disorders) | 11
Hypotension (Vascular disorders) | 12
Lymphoedema (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 2
Superior vena cava syndrome (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Hepatobiliary disease (Hepatobiliary disorders) | 3
Respiratory tract infection (Infections and infestations) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Parosmia (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2012-04-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT01597258/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT01597258/SAP_001.pdf